CLINICAL TRIAL: NCT02095028
Title: Effects of Dietary and Lifestyle Interventions in Obese Pregnant Women From the First Trimester on Gestational Weight Gain and Pregnancy Outcomes
Brief Title: Dietary and Lifestyle Interventions in Obese Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Guanghui Li, Associate Professor, MD,PhD, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011-2011-02; 201002013 (Other: Health industry special funds for Public Benefit)
Record Dates: First submitted 2014-03-19; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Obesity; Weight Gain; Lifestyle; Pregnancy Related
MeSH Terms: conditions — Obesity; Weight Gain | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary and lifestyle intervention (Experimental): Intervention group:Based on standard care,intensive dietary and lifestyle intervention was provided. Initiated from the first trimester to delivery,every 2-4 weeks follow-up
  Interventions: Behavioral: Dietary and lifestyle intervention
- Standard care group (No Intervention): Standard care group:Participants received one group session in which prenatal general dietary, nutrition guideline, physical activity and recommendation for gestational weight gain introduced by a registered dietitian in 1.5hours.Participants received their regularly scheduled visits without additional dietary and lifestyle follow-up and guidance.

INTERVENTIONS:
Behavioral: Dietary and lifestyle intervention — participants in the intervention group were provided with an individualized dietary intake protocol. Patients received a diet of not fewer than 1500 calories per day in the first trimester and not fewer than 1800 calories per day after 13wks of gestation.
  Arms: Dietary and lifestyle intervention

SUMMARY:
Background: Maternal obesity is associated with higher risks of adverse maternal and fetal complications, but the effects of dietary and lifestyle interventions on gestational weight gain(GWG) and pregnancy outcomes in obese pregnant women are unclear.

Objective: This study examined whether intensive dietary and lifestyle interventions initiated in the early pregnancy could decrease GWG, and prevent relevant adverse pregnancy outcomes in Chinese obese pregnant women.

Design:A randomized controlled trial in obese pregnant women was performed at 6-12 weeks of gestation.The sample size was estimated using GWG reduction as the primary outcome variable. The investigators pilot study (data not published) showed the gestational weight gain was 12.73±5.97 for obese women. Assuming intervention may result in 25% (3.1825g) reduction in GWG, the estimated sample size with 90% power and type I error of 0.05 was 114 women in intervention group and 57 in control group. Adjusting for 15% refusal or loss to follow up during pregnancy, the total sample size required was 136 women in intervention group and 68 in control group(standard care group). Participants were randomly assigned to the control or the intervention group. The intervention focused on restricting energy intake combined with behavioral lifestyle modification through participation in group sessions and individual counseling. The primary outcomes were gestational weight gain (GWG) and secondary outcomes were the incidence of gestational diabetes mellitus (GDM), hypertensive disorders during pregnancy, large-for-gestational-age (LGA) infants, macrosomia and the rate of caesarian section.

Hypothesis:The intensive dietary and lifestyle intervention performed from the first trimester in obese women could decrease total GWG,and perhaps improve relevant pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 6 and 12 weeks of gestation, pre-pregnancy≥28 (kg/m2)
* age ≥18 years, and a singleton pregnancy.

Exclusion Criteria:

* patients with prediabetes and diabetes, hypertension, chronic renal disease, thyroid disorder
* gestational weeks ≥ 13
* age <18 years
* multiple pregnancy
* uterine malformation
* or physical restriction that prevents exercise.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 373 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | From enrollment to delivery (28-34 weeks of gestation)

SECONDARY OUTCOMES:
The incidence of gestational diabetes mellitus | From enrollment to delivery (28-34 weeks of gestation)
The incidence of hypertensive disorders during pregnancy | From enrollment to delivery (28-34 weeks of gestation)
The incidence of large-for-gestational-age infants | From enrollment to delivery(28-34 weeks of gestation)
The incidence of macrosomia infants | From enrollment to delivery (28-34 weeks of gestation)
The rate of caesarian section | From enrollment to delivery(28-34 weeks of gestation)

CONTACTS AND LOCATIONS:
Overall Officials: Guanghui Li, MD,PhD, Principal Investigator — Beijing Obstetrics and Gynecology Hospital
Locations (1):
- Beijing Obstetrics and Gynecology Hospital,Capital Medical University, Beijing, China

REFERENCES:
- [Background] Haslam DW, James WP. Obesity. Lancet. 2005 Oct 1;366(9492):1197-209. doi: 10.1016/S0140-6736(05)67483-1. PMID 16198769
- [Background] Heslehurst N, Rankin J, Wilkinson JR, Summerbell CD. A nationally representative study of maternal obesity in England, UK: trends in incidence and demographic inequalities in 619 323 births, 1989-2007. Int J Obes (Lond). 2010 Mar;34(3):420-8. doi: 10.1038/ijo.2009.250. Epub 2009 Dec 22. PMID 20029373
- [Background] Stothard KJ, Tennant PW, Bell R, Rankin J. Maternal overweight and obesity and the risk of congenital anomalies: a systematic review and meta-analysis. JAMA. 2009 Feb 11;301(6):636-50. doi: 10.1001/jama.2009.113. PMID 19211471
- [Background] Mission JF, Marshall NE, Caughey AB. Obesity in pregnancy: a big problem and getting bigger. Obstet Gynecol Surv. 2013 May;68(5):389-99. doi: 10.1097/OGX.0b013e31828738ce. PMID 23624964
- [Background] Oteng-Ntim E, Varma R, Croker H, Poston L, Doyle P. Lifestyle interventions for overweight and obese pregnant women to improve pregnancy outcome: systematic review and meta-analysis. BMC Med. 2012 May 10;10:47. doi: 10.1186/1741-7015-10-47. PMID 22574949
- [Background] Thangaratinam S, Rogozinska E, Jolly K, Glinkowski S, Roseboom T, Tomlinson JW, Kunz R, Mol BW, Coomarasamy A, Khan KS. Effects of interventions in pregnancy on maternal weight and obstetric outcomes: meta-analysis of randomised evidence. BMJ. 2012 May 16;344:e2088. doi: 10.1136/bmj.e2088. PMID 22596383
- [Background] Guelinckx I, Devlieger R, Mullie P, Vansant G. Effect of lifestyle intervention on dietary habits, physical activity, and gestational weight gain in obese pregnant women: a randomized controlled trial. Am J Clin Nutr. 2010 Feb;91(2):373-80. doi: 10.3945/ajcn.2009.28166. Epub 2009 Dec 2. PMID 19955397
- [Background] Phelan S, Phipps MG, Abrams B, Darroch F, Schaffner A, Wing RR. Randomized trial of a behavioral intervention to prevent excessive gestational weight gain: the Fit for Delivery Study. Am J Clin Nutr. 2011 Apr;93(4):772-9. doi: 10.3945/ajcn.110.005306. Epub 2011 Feb 10. PMID 21310836
- [Background] Kinnunen TI, Pasanen M, Aittasalo M, Fogelholm M, Hilakivi-Clarke L, Weiderpass E, Luoto R. Preventing excessive weight gain during pregnancy - a controlled trial in primary health care. Eur J Clin Nutr. 2007 Jul;61(7):884-91. doi: 10.1038/sj.ejcn.1602602. Epub 2007 Jan 17. PMID 17228348
- [Background] Streuling I, Beyerlein A, von Kries R. Can gestational weight gain be modified by increasing physical activity and diet counseling? A meta-analysis of interventional trials. Am J Clin Nutr. 2010 Oct;92(4):678-87. doi: 10.3945/ajcn.2010.29363. Epub 2010 Jul 28. PMID 20668049
- [Background] Nascimento SL, Surita FG, Parpinelli MA, Siani S, Pinto e Silva JL. The effect of an antenatal physical exercise programme on maternal/perinatal outcomes and quality of life in overweight and obese pregnant women: a randomised clinical trial. BJOG. 2011 Nov;118(12):1455-63. doi: 10.1111/j.1471-0528.2011.03084.x. Epub 2011 Sep 6. PMID 21895947
- [Background] Connor Gorber S, Tremblay M, Moher D, Gorber B. A comparison of direct vs. self-report measures for assessing height, weight and body mass index: a systematic review. Obes Rev. 2007 Jul;8(4):307-26. doi: 10.1111/j.1467-789X.2007.00347.x. PMID 17578381
- [Background] Kiel DW, Dodson EA, Artal R, Boehmer TK, Leet TL. Gestational weight gain and pregnancy outcomes in obese women: how much is enough? Obstet Gynecol. 2007 Oct;110(4):752-8. doi: 10.1097/01.AOG.0000278819.17190.87. PMID 17906005
- [Background] Dodd JM, Crowther CA, Robinson JS. Dietary and lifestyle interventions to limit weight gain during pregnancy for obese or overweight women: a systematic review. Acta Obstet Gynecol Scand. 2008;87(7):702-6. doi: 10.1080/00016340802061111. PMID 18607830
- [Result] Carreno CA, Clifton RG, Hauth JC, Myatt L, Roberts JM, Spong CY, Varner MW, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Carpenter MW, Sciscione A, Tolosa JE, Saade GR, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Excessive early gestational weight gain and risk of gestational diabetes mellitus in nulliparous women. Obstet Gynecol. 2012 Jun;119(6):1227-33. doi: 10.1097/AOG.0b013e318256cf1a. Erratum In: Obstet Gynecol. 2012 Sep;120(3):710. Saade, George R [added]. PMID 22617588
- [Result] Gibson KS, Waters TP, Catalano PM. Maternal weight gain in women who develop gestational diabetes mellitus. Obstet Gynecol. 2012 Mar;119(3):560-5. doi: 10.1097/AOG.0b013e31824758e0. PMID 22353954
- [Result] Wolff S, Legarth J, Vangsgaard K, Toubro S, Astrup A. A randomized trial of the effects of dietary counseling on gestational weight gain and glucose metabolism in obese pregnant women. Int J Obes (Lond). 2008 Mar;32(3):495-501. doi: 10.1038/sj.ijo.0803710. Epub 2008 Jan 29. PMID 18227847
- [Result] Asbee SM, Jenkins TR, Butler JR, White J, Elliot M, Rutledge A. Preventing excessive weight gain during pregnancy through dietary and lifestyle counseling: a randomized controlled trial. Obstet Gynecol. 2009 Feb;113(2 Pt 1):305-12. doi: 10.1097/AOG.0b013e318195baef. PMID 19155899
- [Result] Thornton YS, Smarkola C, Kopacz SM, Ishoof SB. Perinatal outcomes in nutritionally monitored obese pregnant women: a randomized clinical trial. J Natl Med Assoc. 2009 Jun;101(6):569-77. doi: 10.1016/s0027-9684(15)30942-1. PMID 19585925
- [Result] Luoto R, Kinnunen TI, Aittasalo M, Kolu P, Raitanen J, Ojala K, Mansikkamaki K, Lamberg S, Vasankari T, Komulainen T, Tulokas S. Primary prevention of gestational diabetes mellitus and large-for-gestational-age newborns by lifestyle counseling: a cluster-randomized controlled trial. PLoS Med. 2011 May;8(5):e1001036. doi: 10.1371/journal.pmed.1001036. Epub 2011 May 17. PMID 21610860